CLINICAL TRIAL: NCT03740165
Title: A Randomized Phase 3, Double-Blind Study of Chemotherapy With or Without Pembrolizumab Followed by Maintenance With Olaparib or Placebo for the First-Line Treatment of BRCA Non-mutated Advanced Epithelial Ovarian Cancer (EOC) (KEYLYNK-001 / ENGOT-ov43 / GOG-3036)
Brief Title: Study of Chemotherapy With Pembrolizumab (MK-3475) Followed by Maintenance With Olaparib (MK-7339) for the First-Line Treatment of Women With BRCA Non-mutated Advanced Epithelial Ovarian Cancer (EOC) (MK-7339-001/KEYLYNK-001/ENGOT-ov43/GOG-3036)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: European Network of Gynaecological Oncological Trial Groups (ENGOT) (Other); Gynecologic Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7339-001; ENGOT-ov43 (Other: European Network of Gynaecological Oncological Trial Groups (ENGOT)); MK-7339-001 (Other: MSD); KEYLYNK-001 (Other: MSD); 194619 (Registry Identifier: Japic-CTI); GOG-3036 (Other: Gynecologic Oncology Group (GOG)); 2022-502124-52-00 (Registry Identifier: EU CT); U1111-1283-3793 (Registry Identifier: UTN); 2018-001973-25 (EudraCT Number)
Record Dates: First submitted 2018-11-12; First posted 2018-11-14 (Actual); Results first posted 2025-09-12 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-09

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Neoplasms
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1)
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Peritoneal Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Saline Solution; Glucose; Carboplatin; Paclitaxel; olaparib; Bevacizumab; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Carboplatin + Paclitaxel + Pembrolizumab + Olaparib (Experimental): Participants receive carboplatin/paclitaxel via intravenous (IV) infusion for five 3-week cycles PLUS pembrolizumab 200 mg via IV infusion on Day 1 of each 3-week cycle for up to 35 cycles PLUS olaparib 300 mg via oral tablet twice each day (BID), starting with Cycle 7. Participants who experience severe hypersensitivity reaction to paclitaxel or an AE requiring discontinuation of paclitaxel may receive docetaxel (75 mg/m^2 Q3W) plus carboplatin AUC 5 Q3W after Sponsor consultation. Participants may also receive bevacizumab via IV infusion on Day 1 of each 3-week cycle at the Investigator's discretion.
  Interventions: Biological: Pembrolizumab; Drug: Carboplatin; Drug: Paclitaxel; Drug: Olaparib; Biological: Bevacizumab; Drug: Docetaxel
- Carboplatin + Paclitaxel + Pembrolizumab (Experimental): Participants receive carboplatin/paclitaxel via IV infusion for five 3-week cycles starting in Cycle 1 PLUS pembrolizumab 200 mg via IV infusion on Day 1 of each 3-week cycle for up to 35 cycles PLUS placebo for olaparib via oral tablet BID, starting with Cycle 7. Participants who experience severe hypersensitivity reaction to paclitaxel or an AE requiring discontinuation of paclitaxel may receive docetaxel (75 mg/m^2 Q3W) plus carboplatin AUC 5 Q3W after Sponsor consultation. Participants may also receive bevacizumab via IV infusion on Day 1 of each 3-week cycle at the Investigator's discretion.
  Interventions: Biological: Pembrolizumab; Drug: Carboplatin; Drug: Paclitaxel; Drug: Placebo for olaparib; Biological: Bevacizumab; Drug: Docetaxel
- Carboplatin + Paclitaxel (Active Comparator): Participants receive carboplatin/paclitaxel via IV infusion for five 3-week cycles PLUS placebo for pembrolizumab (normal saline or dextrose) via IV infusion on Day 1 of each 3-week cycle for up to 35 cycles PLUS placebo for olaparib via oral tablet BID, starting with Cycle 7. Participants who experience severe hypersensitivity reaction to paclitaxel or an AE requiring discontinuation of paclitaxel may receive docetaxel (75 mg/m^2 Q3W) plus carboplatin AUC 5 Q3W after Sponsor consultation. Participants may also receive bevacizumab via IV infusion on Day 1 of each 3-week cycle at the Investigator's discretion.
  Interventions: Drug: Placebo for pembrolizumab; Drug: Carboplatin; Drug: Paclitaxel; Drug: Placebo for olaparib; Biological: Bevacizumab; Drug: Docetaxel

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®
  Arms: Carboplatin + Paclitaxel + Pembrolizumab; Carboplatin + Paclitaxel + Pembrolizumab + Olaparib
Drug: Placebo for pembrolizumab — IV infusion
  Other Names: normal saline or dextrose
  Arms: Carboplatin + Paclitaxel
Drug: Carboplatin — IV infusion
  Other Names: PARAPLATIN®
Drug: Paclitaxel — IV infusion
  Other Names: TAXOL®
Drug: Olaparib — Oral tablet
  Other Names: MK-7339; LYNPARZA®
  Arms: Carboplatin + Paclitaxel + Pembrolizumab + Olaparib
Drug: Placebo for olaparib — Oral tablet
  Arms: Carboplatin + Paclitaxel; Carboplatin + Paclitaxel + Pembrolizumab
Biological: Bevacizumab — IV infusion
  Other Names: AVASTIN®
Drug: Docetaxel — IV infusion

SUMMARY:
The purpose of this study is to assess the efficacy and safety of treatment with carboplatin/paclitaxel* PLUS pembrolizumab (MK-3475) and maintenance olaparib (MK-7339) in women with epithelial ovarian cancer (EOC), fallopian tube cancer, or primary peritoneal cancer.

The primary study hypotheses are that the combination of pembrolizumab plus carboplatin/paclitaxel* followed by continued pembrolizumab and maintenance olaparib is superior to carboplatin/paclitaxel alone with respect to Progression Free Survival (PFS) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) in participants with programmed death-ligand 1 (PD-L1) positive tumors (Combined Positive Score [CPS]≥10) and in all participants, and that the combination of pembrolizumab plus carboplatin/paclitaxel followed by continued pembrolizumab is superior to carboplatin/paclitaxel alone with respect to PFS per RECIST 1.1 in participants with PD-L1 positive tumors (CPS≥10) and in all participants.

DETAILED DESCRIPTION:
Following a lead-in period during which all participants receive a single 3-week cycle of carboplatin/paclitaxel*, participants will be randomly assigned in to one of three treatment arms, and will receive carboplatin/paclitaxel* for 5 cycles plus:

* Pembrolizumab + Olaparib
* Pembrolizumab + Placebo for Olaparib
* Placebo for Pembrolizumab + Placebo for Olaparib

  * At Investigator's discretion and prior to participant randomization, one of the following carboplatin/paclitaxel regimens is to be selected:

    1. up to 5 cycles of carboplatin Area Under the Curve (AUC)5 or AUC6 AND paclitaxel 175 mg/m^2 on Day 1 of each 3-week cycle
    2. up to 5 cycles of carboplatin AUC5 or AUC6 on Day 1 of each 3-week cycle AND paclitaxel 80 mg/m^2 on Days 1, 8 and 15 of each 3-week cycle; or
    3. up to 5 cycles of carboplatin AUC2 or AUC2.7 AND paclitaxel 60 mg/m^2 on Days 1, 8 and 15 of each 3-week cycle.

Docetaxel may be considered for participants who experience either a severe hypersensitivity reaction to paclitaxel or an AE requiring discontinuation of paclitaxel only after consultation with the Sponsor. The recommended dose as determined by the Scottish Gynaecological Cancer Trials Group is Docetaxel 75 mg/m^2 Q3W plus carboplatin AUC 5 Q3W.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically confirmed International Federation of Gynecology and Obstetrics (FIGO) Stage III or Stage IV EOC (high-grade predominantly serous, endometrioid (any grade), carcinosarcoma, mixed mullerian with high-grade serous component, clear cell, or low-grade serous OC), primary peritoneal cancer, or fallopian tube cancer
* Has just completed primary debulking surgery or is eligible for primary debulking surgery or is a potential candidate for interval debulking surgery
* Is a candidate for carboplatin and paclitaxel chemotherapy, to be administered in the adjuvant or neoadjuvant setting
* Candidates for neoadjuvant chemotherapy, has a cancer antigen 125 (CA-125) (kilounits/L):carcinoembryonic antigen (CEA; ng/mL) ratio greater than or equal to 25
* Is able to provide a newly obtained core or excisional biopsy of a tumor lesion for prospective testing of BRCA1/2 and Programmed Cell Death-Ligand 1 (PD-L1) tumor markers status prior to randomization
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1, as assessed within 7 days prior to initiating chemotherapy in the lead-in period and within 3 days prior to Day 1 of Cycle 1
* Female participants are not pregnant, not breastfeeding, and at least 1 of the following conditions applies: a.) Not a woman of childbearing potential (WOCBP) OR b.) Is a WOCBP and using a contraceptive method that is highly effective, with low user dependency, or be abstinent from heterosexual intercourse as their preferred and usual lifestyle, during the Treatment Period and for at least 120 days following the last dose of pembrolizumab (or pembrolizumab placebo) and bevacizumab (if administered), at least 180 days following the last dose of olaparib (or olaparib placebo), and at least 210 days following the last dose of chemotherapy and agrees not to donate eggs (ova, oocytes) to others or freeze/store for her own use for the purpose of reproduction during this period. The investigator should evaluate the potential for contraceptive method failure in relationship to the first dose of study treatment. A WOCBP must have a negative highly sensitive pregnancy test within either 24 hours (urine) or 72 hours (serum) before the first dose of study treatment. If a urine test cannot be confirmed as negative, a serum pregnancy test is required. The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy. Contraceptive use by women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies
* Has adequate organ function

Exclusion Criteria:

* Has mucinous, germ cell, or borderline tumor of the ovary
* Has a known or suspected deleterious mutation (germline or somatic) in either BRCA1 or BRCA2
* Has a history of non-infectious pneumonitis that required treatment with steroids or currently has pneumonitis
* Has either myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) or has features suggestive of MDS/AML
* Has a known additional malignancy that is progressing or has required active treatment in the last 3 years Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. ductal carcinoma in situ, cervical carcinoma in situ) that has undergone potentially curative therapy are not excluded.
* Has ongoing Grade 3 or Grade 4 toxicity, excluding alopecia, following chemotherapy administered during the lead-in period
* Has known active central nervous system metastases and/or carcinomatous meningitis. Participants with brain metastases may participate provided they were previously treated (except with chemotherapy) and are radiologically stable, clinically stable, and no steroids were used for the management of symptoms related to brain metastases within 14 days prior to randomization. Stable brain metastases should be established prior to the first dose of study medication lead-in chemotherapy
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (dosing >10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to randomization
* Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs) Note: Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
* Has a known history of active tuberculosis (TB; Bacillus Tuberculosis)
* Has an active infection requiring systemic therapy
* Has received colony-stimulating factors (eg, granulocyte colony stimulating factor [G-CSF], granulocyte macrophage colony-stimulating factor [GM-CSF] or recombinant erythropoietin) within 4 weeks prior to receiving chemotherapy during the lead-in period
* Is considered to be of poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection
* Has had surgery to treat borderline tumors, early stage EOC, or early stage fallopian tube cancer <6 months prior to screening
* Has a known history of human immunodeficiency virus (HIV) infection
* Has a known history of hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Testing for hepatitis B or hepatitis C is required at screening only if mandated by local health authority. Note: Participants with a history of hepatitis B but who are HBsAg negative are eligible for the study
* Is either unable to swallow orally administered medication or has a gastrointestinal (GI) disorder affecting absorption (e.g. gastrectomy, partial bowel obstruction, malabsorption)
* Has uncontrolled hypertension
* Has current, clinically relevant bowel obstruction (including sub-occlusive disease), abdominal fistula or GI perforation, related to underlying EOC (for participants receiving bevacizumab)
* Has a history of hemorrhage, hemoptysis or active GI bleeding within 6 months prior to randomization (for participants receiving bevacizumab)
* Is a WOCBP who has a positive urine pregnancy test within 72 hours before the first dose of chemotherapy in the lead-in period and within 72 hours prior to Day 1 of Cycle 1, is pregnant or breastfeeding, or is expecting to conceive children within the projected duration of the study, starting with screening through 120 days following the last dose of pembrolizumab (or pembrolizumab placebo) and bevacizumab (if administered), at least 180 days following the last dose of olaparib (or olaparib placebo), and at least 210 days following the last dose of chemotherapy
* Has received prior treatment for any stage of OC, including radiation or systemic anti-cancer therapy (e.g. chemotherapy, hormonal therapy, immunotherapy, investigational therapy)
* Has received prior therapy with an anti-Programmed Cell Death-1 (anti-PD-1), anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g. cytotoxic T lymphocyte antigen-4 [CTLA-4], OX 40, CD137)
* Has received prior therapy with either olaparib or any other poly(adenosine-ribose) polymerase (PARP) inhibitor
* Has intraperitoneal chemotherapy planned or has been administered as first-line therapy
* Has received a live vaccine within 30 days prior to the first dose of study treatment on Day 1 of Cycle 1
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab, olaparib, carboplatin, paclitaxel or bevacizumab (if using) and/or any of their excipients
* Is currently receiving either strong (e.g. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate (eg, ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil) inhibitors of cytochrome P450 (CYP)3A4 that cannot be discontinued for the duration of the study
* Is currently receiving either strong (e.g. phenobarbital, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine, and St John's Wort) or moderate (e.g. bosentan, efavirenz, modafinil) inducers of CYP3A4 that cannot be discontinued for the duration of the study
* Is currently participating or has participated in a study of an investigational agent or has used an investigational device within 4 weeks (28 days) of starting chemotherapy in the Lead-in Period
* Has resting electrocardiogram (ECG) indicating uncontrolled, potentially reversible cardiac conditions or participant has congenital long QT syndrome
* Has had an allogenic tissue/solid organ transplant, has received previous allogenic bone-marrow transplant, or has received double umbilical cord transplantation
* Either has had major surgery within 3 weeks of randomization or has not recovered from any effects of any major surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1367 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2026-05-29 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (227):
- United States (43):
  - University of Alabama at Birmingham (UAB) ( Site 0036), Birmingham, Alabama
  - University of Arizona Cancer Center ( Site 0074), Tucson, Arizona
  - Disney Family Cancer Center ( Site 0042), Burbank, California
  - Kaiser Permanente Oncology Clinical Trial -Oakland ( Site 0077), Oakland, California
  - Kaiser Permanente Oncology Clinical Trials-Roseville ( Site 0084), Roseville, California
  - Kaiser Permanente Oncology Clinical Trials-Sacramento ( Site 0083), Sacramento, California
  - Kaiser Permanente Oncology Clinical Trial - San Francisco ( Site 0078), San Francisco, California
  - Kaiser Permanente Oncology Clinical Trial - Santa Clara ( Site 0079), Santa Clara, California
  - Kaiser Permanente N. CA Regional Oncology Clinical Trials ( Site 0008), Vallejo, California
  - Kaiser Permanente Oncology Clinical Trial - Walnut Creek ( Site 0080), Walnut Creek, California
  - Smilow Cancer Center at Yale-New Haven ( Site 0057), New Haven, Connecticut
  - Sarasota Memorial Hospital ( Site 0023), Sarasota, Florida
  - Emory School of Medicine ( Site 0053), Atlanta, Georgia
  - Northeast Georgia Medical Center ( Site 0029), Gainesville, Georgia
  - Memorial Health University Medical Center ( Site 0011), Savannah, Georgia
  - Rush University Medical Center ( Site 0019), Chicago, Illinois
  - University of Chicago ( Site 0049), Chicago, Illinois
  - Dr. Sudarshan K. Sharma, LTD ( Site 0061), Hinsdale, Illinois
  - Saint Vincent Hospital and Health Center ( Site 0012), Indianapolis, Indiana
  - University of Iowa Hospital and Clinics ( Site 0005), Iowa City, Iowa
  - University of Kentucky ( Site 0045), Lexington, Kentucky
  - Weinberg Cancer Institute at Franklin Square ( Site 0035), Baltimore, Maryland
  - Saint Dominic - Jackson Memorial Hospital ( Site 0072), Jackson, Mississippi
  - Washington University - School of Medicine ( Site 0062), St Louis, Missouri
  - Nebraska Methodist Hospital ( Site 0063), Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center ( Site 0024), Lebanon, New Hampshire
  - MD Anderson Cancer Center at Cooper ( Site 0067), Camden, New Jersey
  - Holy Name Medical Center ( Site 0037), Teaneck, New Jersey
  - Northwell Health- Monter Cancer Center ( Site 0075), Lake Success, New York
  - Sanford Roger Maris Cancer Center ( Site 0082), Fargo, North Dakota
  - Miami Valley Hospital [Dayton, OH] ( Site 0073), Centerville, Ohio
  - Oncology/Hematology Care Clinical Trials, LLC ( Site 8001), Cincinnati, Ohio
  - The Bing Cancer Center ( Site 0044), Columbus, Ohio
  - OSU Wexner Medical Center ( Site 0076), Hilliard, Ohio
  - Women and Infants Hospital [Providence, RI] ( Site 0039), Providence, Rhode Island
  - Sanford Gynecology Oncology ( Site 0004), Sioux Falls, South Dakota
  - Texas Oncology, P.A. - Bedford ( Site 8005), Bedford, Texas
  - Texas Oncology-Dallas Presbyterian Hospital ( Site 8004), Dallas, Texas
  - Parkland Hospital ( Site 0081), Dallas, Texas
  - UT Southwestern Medical Center ( Site 0046), Dallas, Texas
  - Texas Oncology, P.A. Texas Oncology-Tyler ( Site 8006), Tyler, Texas
  - Virginia Cancer Specialists, PC ( Site 8003), Gainesville, Virginia
  - MEDICAL COLLEGE OF WISCONSIN ( Site 0064), Milwaukee, Wisconsin
- Australia (5):
  - St George Hospital ( Site 2207), Kogarah, New South Wales
  - Cairns and Hinterland Hospital and Health Service ( Site 2201), Cairns, Queensland
  - Ballarat Health Services ( Site 2202), Ballarat, Victoria
  - Monash Health ( Site 2204), Clayton, Victoria
  - Sunshine Hospital. ( Site 2205), St Albans, Victoria
- Belgium (9):
  - Imelda Ziekenhuis Bonheiden ( Site 0301), Bonheiden, Antwerpen
  - UZ Leuven Campus Gasthuisberg ( Site 0306), Leuven, Antwerpen
  - Cliniques Universitaires Saint-Luc ( Site 0312), Brussels, Bruxelles-Capitale, Region de
  - Grand Hopital de Charleroi ( Site 0302), Charleroi, Hainaut
  - CHU de Liege ( Site 0310), Liège, Liege
  - Jessa Ziekenhuis ( Site 0309), Hasselt, Limburg
  - Centre Hospitalier de l'Ardenne ( Site 0303), Libramont, Luxembourg
  - AZ Maria Middelares Gent ( Site 0300), Ghent, Oost-Vlaanderen
  - UZ Gent ( Site 0307), Ghent, Oost-Vlaanderen
- Brazil (10):
  - Instituto do Cancer do Ceara ( Site 2707), Fortaleza, Ceará
  - Hospital Araujo Jorge Associacao de Combate ao Cancer de Goias ( Site 2708), Goiânia, Goiás
  - Hospital Erasto Gaertner ( Site 2716), Curitiba, Paraná
  - Hospital de Caridade de Ijui ( Site 2712), Ijuí, Rio Grande do Sul
  - Hospital Bruno Born ( Site 2704), Lajeado, Rio Grande do Sul
  - Hospital Nossa Senhora Da Conceicao ( Site 2703), Porto Alegre, Rio Grande do Sul
  - Instituto Nacional de Cancer Hospital do Cancer II ( Site 2700), Rio de Janeiro
  - Instituto do Cancer do Estado de Sao Paulo - ICESP ( Site 2714), São Paulo
  - Clinica de Pesquisas e Ctro de Estudos Onc. Ginecol. e Mamaria Ltda ( Site 2706), São Paulo
  - Real e Benemerita Associacao Portuguesa de Beneficencia ( Site 2710), São Paulo
- Canada (8):
  - Tom Baker Cancer Centre ( Site 0200), Calgary, Alberta
  - Kingston Health Sciences Centre ( Site 0207), Kingston, Ontario
  - The Credit Valley Hospital ( Site 0206), Mississauga, Ontario
  - Princess Margaret Hospital.. ( Site 0202), Toronto, Ontario
  - CIUSSS du Saguenay-Lac-St-Jean ( Site 0218), Chicoutimi, Quebec
  - CIUSSS de l Est de L Ile de Montreal - Hopital Maisonneuve-Rosemont ( Site 0219), Montreal, Quebec
  - Centre Hospitalier de l Universite de Montreal - CHUM ( Site 0208), Montreal, Quebec
  - Royal Victoria Hospital McGill University Health Centre ( Site 0211), Montreal, Quebec
- Chile (8):
  - Fundacion Arturo Lopez Perez FALP ( Site 2800), Santiago, Region M. de Santiago
  - Sociedad Oncovida S.A. ( Site 2807), Santiago, Region M. de Santiago
  - Iram Cancer Research ( Site 2809), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile ( Site 2805), Santiago, Region M. de Santiago
  - Centro Investigación del Cáncer James Lind ( Site 2810), Temuco, Región de la Araucanía
  - Centro de Investigacion y desarrollo Oncologico SpA - CIDO SpA ( Site 2808), Temuco, Región de la Araucanía
  - Oncocentro ( Site 2801), Viña del Mar, Región de Valparaíso
  - Centro Oncologico Antofagasta ( Site 2804), Antofagasta
- Colombia (7):
  - Biomelab S A S ( Site 2900), Barranquilla, Atlántico
  - Instituto Nacional de Cancerologia E.S.E ( Site 2910), Bogotá, Bogota D.C.
  - Clinica Colsanitas S.A. Sede Clinica Universitaria Colombia ( Site 2912), Bogotá, Bogota D.C.
  - Sociedad de Oncología Y Hematología del Cesar S.A.S. ( Site 2913), Valledupar, Cesar Department
  - Oncomedica S.A. ( Site 2911), Montería, Departamento de Córdoba
  - Centro Medico Imbanaco de Cali S.A ( Site 2909), Cali, Valle del Cauca Department
  - Hemato Oncologos S.A. ( Site 2906), Cali, Valle del Cauca Department
- Czechia (5):
  - Fakultni nemocnice Brno ( Site 0404), Brno, Brno-mesto
  - Fakultni nemocnice Ostrava ( Site 0403), Ostrava-Poruba, Moravskoslezský kraj
  - Vseobecna fakultni nemocnice v Praze ( Site 0400), Prague, Praha, Hlavni Mesto
  - Nemocnice Na Bulovce ( Site 0401), Prague, Praha, Hlavni Mesto
  - Fakultni nemocnice Olomouc ( Site 0402), Olomouc
- France (9):
  - Hopital Prive Jean Mermoz ( Site 0607), Lyon, Auvergne
  - Centre Paul Strauss ( Site 0615), Strasbourg, Bas-Rhin
  - Hopital de la Timone ( Site 0617), Marseille, Bouches-du-Rhone
  - CHU de Brest -Site Hopital Morvan ( Site 0616), Brest, Brittany Region
  - Institut de Cancerologie du Gard - CHU Caremeau ( Site 0610), Nîmes, Gard
  - Centre D Oncologie de Gentilly ( Site 0609), Nancy, Meurthe-et-Moselle
  - Institut de Cancerologie Lucien Neuwirth ( Site 0613), Saint-Priest-en-Jarez, Pays de la Loire Region
  - Institut Gustave Roussy ( Site 0600), Villejuif, Val-de-Marne
  - Hopital Tenon ( Site 0612), Paris
- Germany (12):
  - Marienhospital Stuttgart Vincenz von Paul Kliniken gGmbH ( Site 0707), Stuttgart, Baden-Wurttemberg
  - Klinikum Rechts der Isar. Technischen Universitaet Muenchen ( Site 0710), Munich, Bavaria
  - Uniklinik RWTH Aachen ( Site 0718), Aachen, North Rhine-Westphalia
  - Gynaekologisches Zentrum ( Site 0712), Bonn, North Rhine-Westphalia
  - Klinikum Dortmund gGmbH ( Site 0717), Dortmund, North Rhine-Westphalia
  - Universitaetsklinikum Duesseldorf ( Site 0704), Düsseldorf, North Rhine-Westphalia
  - HELIOS Klinikum Krefeld ( Site 0715), Krefeld, North Rhine-Westphalia
  - Universitaetsklinikum Muenster ( Site 0720), Münster, North Rhine-Westphalia
  - Caritas Klinikum Saarbruecken St. Theresia ( Site 0702), Saarbrücken, Saarland
  - Klinikum Chemnitz gGmbH ( Site 0711), Chemnitz, Saxony
  - Staedtisches Krankenhaus Kiel GmbH ( Site 0709), Kiel, Schleswig-Holstein
  - Charite Campus Virchow-Klinikum - CVK ( Site 0700), Berlin
- Hungary (5):
  - Pecsi Tudomanyegyetem Klinikai Kozpont ( Site 0805), Pécs, Baranya
  - Borsod-Abauj-Zemplen Megyei Korhaz es Egyetemi Oktato Korhaz ( Site 0802), Miskolc, Borsod-Abauj Zemplen county
  - Orszagos Onkologiai Intezet ( Site 0800), Budapest
  - Uzsoki Utcai Korhaz ( Site 0803), Budapest
  - Debreceni Egyetem Klinikai Kozpont ( Site 0801), Debrecen
- Israel (9):
  - Soroka Medical Center ( Site 1006), Beersheba
  - Hillel Yaffe Medical Center ( Site 1011), Hadera
  - Carmel Medical Center ( Site 1007), Haifa
  - Rambam Medical Center ( Site 1002), Haifa
  - Edith Wolfson Medical Center ( Site 1003), Holon
  - Shaare Zedek Medical Center ( Site 1005), Jerusalem
  - Rabin Medical Center ( Site 1004), Petah Tikva
  - Chaim Sheba Medical Center ( Site 1000), Ramat Gan
  - Sourasky Medical Center ( Site 1001), Tel Aviv
- Italy (13):
  - IRCCS Giovanni Paolo II. Ospedale Oncologico ( Site 1108), Bari, Abruzzo
  - Istituto Europeo di Oncologia ( Site 1100), Milan, Lombardy
  - A.O.U. Citta della Salute e della Scienza di Torino ( Site 1104), Turin, Piedmont
  - Istituto Oncologico Veneto IRCCS ( Site 1113), Padua, Veneto
  - Sacro Cuore di Gesu Fatebenefratelli ( Site 1112), Benevento
  - Ospedale Cannizzaro ( Site 1110), Catania
  - ASST Lecco. Ospedale A. Manzoni ( Site 1101), Lecco
  - Fondazione IRCCS Istituto Nazionale dei Tumori di Milano ( Site 1115), Milan
  - A.O.U. Federico II di Napoli ( Site 1107), Napoli
  - Azienda Ospedaliera Policlinico Umberto I ( Site 1111), Roma
  - Policlinico Universitario Gemelli ( Site 1105), Roma
  - Presidio Ospedaliero Santa Chiara ( Site 1109), Trento
  - A.O. Univ. S. M. della Misericordia ( Site 1114), Udine
- Japan (16):
  - National Cancer Center Hospital East ( Site 2602), Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center ( Site 2601), Matsuyama, Ehime
  - Ehime University Hospital ( Site 2600), Tōon, Ehime
  - Gunma Prefectural Cancer Center ( Site 2609), Ōta, Gunma
  - Hokkaido University Hospital ( Site 2607), Sapporo, Hokkaido
  - Iwate Medical University Hospital ( Site 2606), Shiwa-gun, Iwate
  - St. Marianna University School of Medicine Hospital ( Site 2613), Kawasaki, Kanagawa
  - University of the Ryukyus Hospital ( Site 2616), Nakagami-gun, Okinawa
  - Saitama Medical University International Medical Center ( Site 2604), Hidaka, Saitama
  - Saitama Cancer Center ( Site 2614), Kitaadachi-gun, Saitama
  - National Defense Medical College Hospital ( Site 2608), Tokorozawa, Saitama
  - Kyorin University Hospital ( Site 2610), Mitaka, Tokyo
  - Kagoshima City Hospital ( Site 2612), Kagoshima
  - Niigata Cancer Center Hospital ( Site 2618), Niigata
  - Osaka International Cancer Institute ( Site 2617), Osaka
  - National Cancer Center Hospital ( Site 2605), Tokyo
- Poland (6):
  - Szpital Kliniczny im. Przemienienia Panskiego Uniwersytetu Medycznego im. K. Marcinkowskiego w Pozna, Poznan, Greater Poland Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy w Warszawie (, Warsaw, Masovian Voivodeship
  - Bialostockie Centrum Onkologii ( Site 1412), Bialystok, Podlaskie Voivodeship
  - Szpitale Pomorskie Sp. z o.o. ( Site 1407), Gdynia, Pomeranian Voivodeship
  - Narodowy Instytut Onkologii - Oddzial w Gliwicach ( Site 1406), Gliwice, Silesian Voivodeship
  - Swietokrzyskie Centrum Onkologii SPZOZ ( Site 1410), Kielce, Świętokrzyskie Voivodeship
- Russia (9):
  - Arkhangelsk Clinical Oncological Dispensary ( Site 1508), Arkhangelsk, Arkhangelskaya oblast
  - Republican Clinical Oncology Dispensary of Republic of Bashkortostan ( Site 1507), Ufa, Baskortostan, Respublika
  - A. Tsyb Medical Radiological Research Center ( Site 1513), Obninsk, Kaluzskaja Oblast
  - FSBI National Medical Oncology Research Center n.a. N.N. Blokhina ( Site 1500), Moscow, Moscow
  - FSCC of Special Types of Med. Care and Technologies ( Site 1503), Moscow, Moscow
  - Medical Rehabilitation Center ( Site 1502), Moscow, Moscow
  - National Medical Research Center of Oncology N.A. N.N. Petrov ( Site 1504), Saint Petersburg, Sankt-Peterburg
  - City Clinical Oncology Center ( Site 1505), Saint Petersburg, Sankt-Peterburg
  - Republican Clinical Oncology Dispensary of Tatarstan MoH ( Site 1509), Kazan', Tatarstan, Respublika
- South Africa (12):
  - Cancer Care Langenhoven Drive Oncology Centre ( Site 1701), Port Elizabeth, Eastern Cape
  - Groote Schuur Hospital ( Site 1704), Cape Town, Gauteng
  - Wits Clinical Research ( Site 1702), Johannesburg, Gauteng
  - Department of Medical Oncology ( Site 1703), Pretoria, Gauteng
  - Curo Oncology ( Site 1710), Pretoria, Gauteng
  - Wilgers Oncology Centre ( Site 1705), Pretoria, Gauteng
  - Little Company of Mary Hospital ( Site 1700), Pretoria, Gauteng
  - Sandton Oncology Medical Group PTY LTD ( Site 1712), Sandton, Gauteng
  - The Oncology Centre ( Site 1709), Durban, KwaZulu-Natal
  - Cancercare ( Site 1706), Cape Town, Western Cape
  - Outeniqua Cancercare Oncology Unit ( Site 1708), George, Western Cape
  - Cape Town Oncology Trials Pty Ltd ( Site 1707), Kraaifontein, Western Cape
- South Korea (5):
  - Seoul National University Bundang Hospital ( Site 2404), Seongnam-si, Kyonggi-do
  - Seoul National University Hospital ( Site 2403), Seoul
  - Severance Hospital Yonsei University Health System ( Site 2400), Seoul
  - Asan Medical Center ( Site 2402), Seoul
  - Samsung Medical Center ( Site 2401), Seoul
- Spain (11):
  - Instituto Catalan de Oncologia ICO - Hospital Duran i Reynals ( Site 1603), L'Hospitalet de Llobregat, Barcelona
  - Xarxa Assistencial Universitaria Manresa ( Site 1605), Manresa, Barcelona
  - Hospital de Terrassa ( Site 1606), Terrassa, Barcelona
  - Hospital Universitario de Donostia ( Site 1602), Donostia / San Sebastian, Gipuzkoa
  - Complejo Hospitalario Universitario A Coruna. CHUAC ( Site 1608), A Coruña, La Coruna
  - Instituto Valenciano de Oncologia ( Site 1601), Valencia, Valenciana, Comunitat
  - Hospital General Universitario de Valencia ( Site 1610), Valencia, Valenciana, Comunitat
  - Hospital Provincial San Pedro de Alcantara ( Site 1607), Cáceres
  - Hospital Universitario Lucus Augusti ( Site 1609), Lugo
  - Clinica Universitaria de Navarra ( Site 1600), Madrid
  - Hospital Universitario Virgen del Rocio ( Site 1604), Seville
- Taiwan (8):
  - Changhua Christian Hospital ( Site 2507), Changhua
  - China Medical University Hospital ( Site 2506), Taichung
  - Taichung Veterans General Hospital ( Site 2510), Taichung
  - National Cheng Kung University Hospital ( Site 2508), Tainan
  - National Taiwan University Hospital ( Site 2502), Taipei
  - MacKay Memorial Hospital ( Site 2500), Taipei
  - Taipei Veterans General Hospital ( Site 2503), Taipei
  - Linkou Chang Gung Memorial Hospital ( Site 2501), Taoyuan District
- Turkey (Türkiye) (9):
  - Istanbul Acibadem University Atakent Hospital ( Site 1902), Küçükçekmece, Istanbul
  - Etlik Zubeyde Hanim Kadin Hastaliklari Egitim ve Arastirma Hastanesi ( Site 1903), Ankara
  - Ankara UTF Cebeci Arastırma ve Uygulama Hastanesi ( Site 1905), Ankara
  - Akdeniz Universitesi Tıp Fakultesi ( Site 1901), Antalya
  - Uludag Universitesi Tip Fakultesi ( Site 1904), Bursa
  - Istanbul Universitesi Istanbul Tip Fakultesi ( Site 1900), Istanbul
  - Bakirkoy Sadi Konuk Egitim ve Arastirma Hastanesi ( Site 1907), Istanbul
  - Medipol Universite Hastanesi ( Site 1909), Istanbul
  - Sakarya Universitesi Tip Fakultesi Hastanesi ( Site 1906), Sakarya
- Ukraine (8):
  - MI Precarpathian Clinical Oncology Center ( Site 2181), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Grigoriev Institute for medical Radiology NAMS of Ukraine ( Site 2180), Kharkiv, Kharkivs’ka Oblast’
  - Municipal non-profit Enterprise Khmelnytskyi Regional Antitu-Gynecological Oncology department, Poli, Khmelnytskyi, Khmelnytskyi Oblast
  - Lviv State Oncology Regional Treatment and Diagnostic Center ( Site 2170), Lviv, Lviv Oblast
  - MI Odessa Regional Oncological Centre ( Site 2121), Odesa, Odesa Oblast
  - RMI - Sumy Regional Clinical Oncology Dispensary ( Site 2191), Sumy, Sumska Oblast
  - Central City Clinical Hospital ( Site 2150), Uzhhorod, Zakarpattia Oblast
  - Kyiv City Clinical Oncological Center ( Site 2140), Kyiv

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26264&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Carboplatin + Paclitaxel + Pembrolizumab + Olaparib | Carboplatin + Paclitaxel + Pembrolizumab | Carboplatin + Paclitaxel
Started | 455 | 458 | 454
Treated | 452 | 456 | 454
Completed | 0 | 0 | 0
Not Completed | 455 | 458 | 454
Not completed — Death | 232 | 242 | 229
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal by Subject | 7 | 4 | 3
Not completed — Ongoing in Study | 216 | 212 | 221

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carboplatin + Paclitaxel + Pembrolizumab + Olaparib | Carboplatin + Paclitaxel + Pembrolizumab | Carboplatin + Paclitaxel | Total
Number analyzed (Participants) | 455 | 458 | 454 | 1367
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.4 (10.6) | 59.8 (11.0) | 59.3 (11.6) | 59.8 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 455 | 458 | 454 | 1367
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 45 | 41 | 45 | 131
  Not Hispanic or Latino | 410 | 415 | 407 | 1232
  Unknown or Not Reported | 0 | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 4 | 0 | 5
  Asian | 77 | 73 | 83 | 233
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 4 | 4 | 15
  White | 360 | 367 | 357 | 1084
  More than one race | 10 | 8 | 9 | 27
  Unknown or Not Reported | 0 | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by the Investigator in Participants With Programmed Death-Ligand 1 (PD-L1) Positive Tumors (Combined Positive Score [CPS]≥10)
Description: PFS is defined as the time from randomization to the first documented progressive disease (PD) per RECIST 1.1 based on Investigator assessment or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions and the unequivocal progression of non-target lesions is also considered PD. The PFS per RECIST 1.1 as assessed by the Investigator will be reported for participants with PD-L1 positive tumors (CPS≥10). PFS was calculated using the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to approximately 67 months
Population: The analysis population includes all randomized participants with CPS≥10. Participants were analyzed in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Carboplatin + Paclitaxel + Pembrolizumab + Olaparib | Carboplatin + Paclitaxel + Pembrolizumab | Carboplatin + Paclitaxel
Number analyzed (Participants) | 229 | 230 | 228
Months | 23.9 [21.0 to 30.2] | 17.3 [15.2 to 19.4] | 15.2 [12.5 to 17.2]
Statistical Analysis 1: Comparison: Carboplatin + Paclitaxel + Pembrolizumab + Olaparib vs Carboplatin + Paclitaxel; Test type: Superiority; p = 0.0002, Log Rank — One-sided p-value based on log-rank test stratified by debulking surgery (planned interval vs R0 following primary vs R1 following primary) and bevacizumab use (Yes vs No); Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.53 to 0.83] — Based on Cox regression model with Efron's method of tie handling; treatment as covariate stratified by debulking surgery (planned interval vs R0 following primary vs R1 following primary) and bevacizumab use (Yes vs No)
Statistical Analysis 2: Comparison: Carboplatin + Paclitaxel + Pembrolizumab vs Carboplatin + Paclitaxel; Test type: Superiority; p = 0.3339, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.77 to 1.19] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: PFS Per RECIST 1.1 as Assessed by the Investigator in All Participants
Description: PFS is defined as the time from randomization to the first documented progressive disease (PD) per RECIST 1.1 based on Investigator assessment or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions and the unequivocal progression of non-target lesions is also considered PD. The PFS per RECIST 1.1 as assessed by the Investigator will be reported for all participants. PFS was calculated using the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to approximately 67 months
Population: The analysis population includes all randomized participants. Participants were analyzed in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Carboplatin + Paclitaxel + Pembrolizumab + Olaparib | Carboplatin + Paclitaxel + Pembrolizumab | Carboplatin + Paclitaxel
Number analyzed (Participants) | 455 | 458 | 454
Months | 22.2 [18.8 to 24.7] | 15.2 [13.6 to 16.4] | 14.6 [12.7 to 16.3]
Statistical Analysis 1: Comparison: Carboplatin + Paclitaxel + Pembrolizumab + Olaparib vs Carboplatin + Paclitaxel; Test type: Superiority; p < 0.0001, Log Rank — One-sided p-value based on log-rank test stratified by debulking surgery (planned interval vs R0 following primary vs R1 following primary), bevacizumab use (Yes vs No), and PD-L1 CPS (<10 vs ≥10); Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.61 to 0.84] — Based on Cox regression model with Efron's method of tie handling; treatment as covariate stratified by debulking surgery (planned interval vs R0 following primary vs R1 following primary), bevacizumab use (Yes vs No), and PD-L1 CPS (<10 vs ≥10)
Statistical Analysis 2: Comparison: Carboplatin + Paclitaxel + Pembrolizumab vs Carboplatin + Paclitaxel; Test type: Superiority; p = 0.5527, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.87 to 1.18] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Overall Survival (OS) in Participants With PD-L1 Positive Tumors (CPS ≥ 10)
Description: OS is defined as the time from the date of randomization to death due to any cause. The OS is reported for all participants with PD-L1 positive tumors (CPS≥10). The OS was calculated using the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to approximately 67 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Carboplatin + Paclitaxel + Pembrolizumab + Olaparib | Carboplatin + Paclitaxel + Pembrolizumab | Carboplatin + Paclitaxel
Number analyzed (Participants) | 229 | 230 | 228
Months | 50.2 [43.9 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event | 56.4 [42.4 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event | 51.6 [41.8 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event
Statistical Analysis 1: Comparison: Carboplatin + Paclitaxel + Pembrolizumab + Olaparib vs Carboplatin + Paclitaxel; Test type: Superiority; p = 0.4314, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.75 to 1.27] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Carboplatin + Paclitaxel + Pembrolizumab vs Carboplatin + Paclitaxel; Test type: Superiority; p = 0.3107, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.72 to 1.22] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: OS in All Participants
Description: OS is defined as the time from the date of randomization to death due to any cause. The OS was calculated using the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to approximately 67 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Carboplatin + Paclitaxel + Pembrolizumab + Olaparib | Carboplatin + Paclitaxel + Pembrolizumab | Carboplatin + Paclitaxel
Number analyzed (Participants) | 455 | 458 | 454
Months | 47.7 [42.3 to 54.9] | 44.2 [38.1 to 52.2] | 47.1 [41.7 to 60.9]
Statistical Analysis 1: Comparison: Carboplatin + Paclitaxel + Pembrolizumab + Olaparib vs Carboplatin + Paclitaxel; Test type: Superiority; p = 0.6716, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.87 to 1.25] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Carboplatin + Paclitaxel + Pembrolizumab vs Carboplatin + Paclitaxel; Test type: Superiority; p = 0.7448, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.89 to 1.27] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: PFS Per RECIST 1.1 as Assessed by Blinded Independent Central Review (BICR) in Participants With PD-L1 Positive Tumors (CPS≥10)
Description: PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1 based on blinded independent central review assessment or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions and the unequivocal progression of non-target lesions is also considered PD. The PFS per RECIST 1.1 as assessed by blinded independent central review will be reported for participants with PD-L1 positive (CPS≥10) tumors (CPS≥10). PFS was calculated using the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to approximately 66 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Carboplatin + Paclitaxel + Pembrolizumab + Olaparib | Carboplatin + Paclitaxel + Pembrolizumab | Carboplatin + Paclitaxel
Number analyzed (Participants) | 229 | 230 | 228
Months | 42.0 [27.2 to 51.9] | 20.3 [17.3 to 27.4] | 22.1 [15.4 to 29.5]
Statistical Analysis 1: Comparison: Carboplatin + Paclitaxel + Pembrolizumab + Olaparib vs Carboplatin + Paclitaxel; Test type: Superiority; p = 0.0012, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.50 to 0.86] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Carboplatin + Paclitaxel + Pembrolizumab vs Carboplatin + Paclitaxel; Test type: Superiority; p = 0.4366, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.75 to 1.27] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: PFS Per RECIST 1.1 as Assessed by BICR in All Participants
Description: PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1 based on blinded independent central review assessment or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions and the unequivocal progression of non-target lesions is also considered PD. The PFS per RECIST 1.1 as assessed by blinded independent central review will be reported for all participants. PFS was calculated using the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to approximately 66 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Carboplatin + Paclitaxel + Pembrolizumab + Olaparib | Carboplatin + Paclitaxel + Pembrolizumab | Carboplatin + Paclitaxel
Number analyzed (Participants) | 455 | 458 | 454
Months | 30.1 [24.0 to 37.3] | 19.0 [16.6 to 22.2] | 20.8 [16.9 to 25.3]
Statistical Analysis 1: Comparison: Carboplatin + Paclitaxel + Pembrolizumab + Olaparib vs Carboplatin + Paclitaxel; Test type: Superiority; p = 0.0008, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.61 to 0.89] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Carboplatin + Paclitaxel + Pembrolizumab vs Carboplatin + Paclitaxel; Test type: Superiority; p = 0.7174, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.88 to 1.27] — [estimate comment as in outcome 2, analysis 1]

7. Secondary Outcome: PFS After Second-line Treatment (PFS2) Following Discontinuation of Study Treatment as Assessed by the Investigator in Participants With PD-L1 Positive Tumors (CPS≥10)
Description: PFS2 is defined as the time from randomization until PD after second-line treatment per RECIST 1.1 based on Investigator assessment, or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions and the unequivocal progression of non-target lesions is also considered PD. The PFS2 per RECIST 1.1 as assessed by the Investigator is reported for participants with PD-L1 positive tumors (CPS≥10). PFS2 was calculated using the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to approximately 67 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Carboplatin + Paclitaxel + Pembrolizumab + Olaparib | Carboplatin + Paclitaxel + Pembrolizumab | Carboplatin + Paclitaxel
Number analyzed (Participants) | 229 | 230 | 228
Months | 41.1 [32.3 to 52.1] | 34.1 [29.0 to 41.2] | 29.9 [25.3 to 37.6]
Statistical Analysis 1: Comparison: Carboplatin + Paclitaxel + Pembrolizumab + Olaparib vs Carboplatin + Paclitaxel; Test type: Superiority; p = 0.0228, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.62 to 1.00] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Carboplatin + Paclitaxel + Pembrolizumab vs Carboplatin + Paclitaxel; Test type: Superiority; p = 0.3935, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.77 to 1.22] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: PFS2 Following Discontinuation of Study Treatment as Assessed by the Investigator in All Participants
Description: PFS2 is defined as the time from randomization until PD after second-line treatment per RECIST 1.1 based on Investigator assessment, or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions and the unequivocal progression of non-target lesions is also considered PD. The PFS2 per RECIST 1.1 as assessed by the Investigator is reported for all participants. PFS2 was calculated using the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to approximately 67 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Carboplatin + Paclitaxel + Pembrolizumab + Olaparib | Carboplatin + Paclitaxel + Pembrolizumab | Carboplatin + Paclitaxel
Number analyzed (Participants) | 455 | 458 | 454
Months | 33.1 [29.9 to 38.5] | 27.8 [26.0 to 32.5] | 28.9 [25.4 to 34.2]
Statistical Analysis 1: Comparison: Carboplatin + Paclitaxel + Pembrolizumab + Olaparib vs Carboplatin + Paclitaxel; Test type: Superiority; p = 0.0573, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.74 to 1.03] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Carboplatin + Paclitaxel + Pembrolizumab vs Carboplatin + Paclitaxel; Test type: Superiority; p = 0.7234, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.89 to 1.23] — [estimate comment as in outcome 2, analysis 1]

9. Secondary Outcome: Change From Baseline in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Global Health Status (Item 29) and Quality of Life (Item 30) (GHS/QoL) Combined Score
Description: The EORTC-QLQ-C30 is a 30-item questionnaire to assess the quality of life of cancer patients. Participant responses to the Global Health Status (GHS) question "How would you rate your overall health during the past week?" (Item 29) and the Quality of Life (QoL) question "How would you rate your overall quality of life during the past week?" (Item 30) were scored on a 7-point scale (1=Very Poor; 7=Excellent). Using linear transformation, raw scores were standardized so scores ranged from 0 to 100; higher score = better outcome. Change from baseline to Week 45 in EORTC QLQ-C30 Items 29 and 30 combined scores was calculated based on a constrained longitudinal data analysis (cLDA) with scores as response variable; covariates for treatment by time interaction and stratification factors (debulking surgery [planned interval vs R0 following primary vs R1 following primary], and bevacizumab use [Yes vs No], and PD-L1 CPS [<10 vs ≥10]).
Time Frame: Baseline and week 45
Population: The analysis population includes all randomized participants who have at least 1 GHS/QoL assessment available and received at least 1 dose of study medication. Participants were analyzed in the treatment group to which they were randomized.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Carboplatin + Paclitaxel + Pembrolizumab + Olaparib | Carboplatin + Paclitaxel + Pembrolizumab | Carboplatin + Paclitaxel
Number analyzed (Participants) | 446 | 455 | 451
Score on a Scale
  cLDA model using Carboplatin+Paclitaxel+Pembrolizumab+Olaparib and Carboplatin+Paclitaxel arms: number analyzed (Participants) | 446 | 0 | 451
  cLDA model using Carboplatin+Paclitaxel+Pembrolizumab+Olaparib and Carboplatin+Paclitaxel arms | 0.45 [-1.62 to 2.52] |  | 0.18 [-1.87 to 2.24]
  cLDA model using Carboplatin+Paclitaxel+Pembrolizumab and Carboplatin+Paclitaxel arms: number analyzed (Participants) | 0 | 455 | 451
  cLDA model using Carboplatin+Paclitaxel+Pembrolizumab and Carboplatin+Paclitaxel arms |  | -0.49 [-2.63 to 1.65] | 0.61 [-1.48 to 2.70]
Statistical Analysis 1: Comparison: Carboplatin + Paclitaxel + Pembrolizumab + Olaparib vs Carboplatin + Paclitaxel; Test type: Superiority; p = 0.8481, t-test, 2 sided; Difference in Least Squares Means (LSM) = 0.26, 95% CI 2-sided [-2.44 to 2.97] — Based on cLDA model with scores as response variable; covariates for treatment by time interaction and stratification factors (debulking surgery [planned interval vs R0 following primary vs R1 following primary], bevacizumab use, and PD-L1 CPS)
Statistical Analysis 2: Comparison: Carboplatin + Paclitaxel + Pembrolizumab vs Carboplatin + Paclitaxel; Test type: Superiority; p = 0.4335, t-test, 2 sided; Difference in LS Means = -1.10, 95% CI 2-sided [-3.87 to 1.66] — [estimate comment as in outcome 9, analysis 1]

10. Secondary Outcome: Mean Change From Baseline in Abdominal and Gastrointestinal (Abdominal/GI) Symptoms Score Using the EORTC Quality of Life Questionnaire-Ovarian Cancer (QLQ-OV28) Abdominal/GI Symptom Scale
Description: Participant responses to 6 questions from the EORTC QoL Questionnaire-Ovarian Cancer (QLQ-OV28) abdominal/GI symptom scale about abdominal pain, bloated feeling in abdomen/stomach, changes in clothing fit, changes in bowel habit, flatulence, and stomach fullness when eating (questions 31-36) were scored on a 4-point scale (1=Not at all; 4=Very much); lower score = better abdominal/GI symptoms. Using linear transformation, raw scores were standardized so that scores ranged from 0 to 100; a lower score indicating a better overall outcome. Change from baseline to Week 45 in EORTC QLQ-OV28 Items 31-36 combined scores was calculated based on a constrained longitudinal data analysis (cLDA) model with scores as response variable; covariates for treatment by time interaction and stratification factors (debulking surgery [planned interval vs R0 following primary vs R1 following primary], and bevacizumab use [Yes vs No], and PD-L1 CPS [<10 vs ≥10]).
Time Frame: Baseline and week 45
Population: The analysis population includes all randomized participants who have at least 1 Abdominal/GI Symptom Scale assessment available and received at least 1 dose of study medication. Participants were analyzed in the treatment group to which they were randomized.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Carboplatin + Paclitaxel + Pembrolizumab + Olaparib | Carboplatin + Paclitaxel + Pembrolizumab | Carboplatin + Paclitaxel
Number analyzed (Participants) | 446 | 454 | 451
Score on a Scale
  cLDA model using Carboplatin+Paclitaxel+Pembrolizumab+Olaparib and Carboplatin+Paclitaxel arms: number analyzed (Participants) | 446 | 0 | 451
  cLDA model using Carboplatin+Paclitaxel+Pembrolizumab+Olaparib and Carboplatin+Paclitaxel arms | -2.63 [-4.40 to -0.85] |  | -2.77 [-4.54 to -1.00]
  cLDA model using Carboplatin+Paclitaxel+Pembrolizumab and Carboplatin+Paclitaxel arms: number analyzed (Participants) | 0 | 454 | 451
  cLDA model using Carboplatin+Paclitaxel+Pembrolizumab and Carboplatin+Paclitaxel arms |  | -2.66 [-4.50 to -0.82] | -2.58 [-4.38 to -0.79]
Statistical Analysis 1: Comparison: Carboplatin + Paclitaxel + Pembrolizumab + Olaparib vs Carboplatin + Paclitaxel; Test type: Superiority; p = 0.9024, t-test, 2 sided; Difference in Least Squares Means (LSM) = 0.14, 95% CI 2-sided [-2.15 to 2.44] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Carboplatin + Paclitaxel + Pembrolizumab vs Carboplatin + Paclitaxel; Test type: Superiority; p = 0.9478, t-test, 2 sided; Difference in Least Squares Means (LSM) = -0.08, 95% CI 2-sided [-2.47 to 2.31] — [estimate comment as in outcome 9, analysis 1]

11. Secondary Outcome: Time to Deterioration (TTD) in European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) Global Health Status (Item 29) and Quality of Life (Item 30) Combined Score
Description: The EORTC-QLQ-C30 is a 30-item questionnaire to assess the quality of life of cancer patients. Participant responses to the Global Health Status (GHS) question "How would you rate your overall health during the past week?" (Item 29) and the Quality of Life (QoL) question "How would you rate your overall quality of life during the past week?" (Item 30) were scored on a 7-point scale (1=Very Poor; 7=Excellent). Using linear transformation, raw scores were standardized so scores ranged from 0 to 100; higher score = better outcome. TTD is defined as the time from the first EORTC QLQ-C30 Items 29 and 30 combined scores to deterioration (defined as ≥10-point decrease in GHS/QoL score from baseline with confirmation under right-censoring rule [the last observation]) or death, whichever occurs first. TTD was calculated using the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to approximately 31 months
Population: The analysis population includes all randomized participants who have at least 1 GHS/QoL assessment available plus a baseline assessment, and received at least 1 dose of study medication. Participants were analyzed in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Carboplatin + Paclitaxel + Pembrolizumab + Olaparib | Carboplatin + Paclitaxel + Pembrolizumab | Carboplatin + Paclitaxel
Number analyzed (Participants) | 420 | 422 | 420
Months | NA [NA to NA] — NA = Median, upper limit, and lower limit not reached at time of data cut-off due to insufficient number of participants with deterioration. | NA [NA to NA] — NA = Median, upper limit, and lower limit not reached at time of data cut-off due to insufficient number of participants with deterioration. | NA [NA to NA] — NA = Median, upper limit, and lower limit not reached at time of data cut-off due to insufficient number of participants with deterioration.
Statistical Analysis 1: Comparison: Carboplatin + Paclitaxel + Pembrolizumab + Olaparib vs Carboplatin + Paclitaxel; Test type: Superiority; p = 0.2644, Log Rank — One-sided p-value based on log-rank test stratified by surgery (planned interval debulking versus R0 following primary debulking versus R1 following primary debulking), bevacizumab use (yes versus no), and PD-L1 status (CPS<10 vs CPS≥10); Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.73 to 1.17] — Based on Cox regression model with Efron's method of tie handling; treatment as covariate stratified by surgery (planned interval vs R0 following primary vs R1 following primary debulking), bevacizumab use (Yes vs No), PD-L1 status (CPS<10 vs CPS≥10)
Statistical Analysis 2: Comparison: Carboplatin + Paclitaxel + Pembrolizumab vs Carboplatin + Paclitaxel; Test type: Superiority; p = 0.1953, Log Rank — [p-value comment as in outcome 11, analysis 1]; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.71 to 1.14] — [estimate comment as in outcome 11, analysis 1]

12. Secondary Outcome: Time to Deterioration (TTD) of Abdominal/GI Symptoms Using EORTC QLQ-OV28
Description: Participant responses to 6 questions from the EORTC QoL Questionnaire-Ovarian Cancer (QLQ-OV28) abdominal/GI symptom scale about abdominal pain, bloated feeling in abdomen/stomach, changes in clothing fit, changes in bowel habit, flatulence, and stomach fullness when eating (questions 31-36) were scored on a 4-point scale (1=Not at all; 4=Very much); lower score = better abdominal/GI symptoms. Using linear transformation, raw scores were standardized so that scores ranged from 0 to 100; a lower score indicating a better overall outcome. TTD is defined as the time from the first EORTC QLQ-OV28 questions 31-36 combined scores to deterioration (defined as ≥10-point decrease in abdominal/GI symptoms score from baseline with confirmation under right-censoring rule [the last observation]) or death, whichever occurs first. TTD was calculated using the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to approximately 31 months
Population: The analysis population includes all randomized participants who have at least 1 Abdominal/GI Symptom Scale assessment available plus a baseline assessment, and received at least 1 dose of study medication. Participants were analyzed in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Carboplatin + Paclitaxel + Pembrolizumab + Olaparib | Carboplatin + Paclitaxel + Pembrolizumab | Carboplatin + Paclitaxel
Number analyzed (Participants) | 416 | 419 | 417
Months | NA [NA to NA] — NA = Median, upper limit, and lower limit not reached at time of data cut-off due to insufficient number of participants with deterioration. | NA [NA to NA] — NA = Median, upper limit, and lower limit not reached at time of data cut-off due to insufficient number of participants with deterioration. | NA [NA to NA] — NA = Median, upper limit, and lower limit not reached at time of data cut-off due to insufficient number of participants with deterioration.
Statistical Analysis 1: Comparison: Carboplatin + Paclitaxel + Pembrolizumab + Olaparib vs Carboplatin + Paclitaxel; Test type: Superiority; p = 0.5188, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.77 to 1.30] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Carboplatin + Paclitaxel + Pembrolizumab vs Carboplatin + Paclitaxel; Test type: Superiority; p = 0.5091, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.77 to 1.30] — [estimate comment as in outcome 2, analysis 1]

13. Secondary Outcome: Time to First Subsequent Anti-cancer Treatment (TFST) in Participants With PD-L1 Positive Tumors (CPS≥10)
Description: TFST is defined as the time from randomization to initiation of first subsequent anti-cancer treatment or death due to any cause, whichever occurs first. The TFST was determined from the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to approximately 67 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Carboplatin + Paclitaxel + Pembrolizumab + Olaparib | Carboplatin + Paclitaxel + Pembrolizumab | Carboplatin + Paclitaxel
Number analyzed (Participants) | 229 | 230 | 228
Months | 29.3 [24.0 to 33.8] | 22.2 [17.7 to 25.4] | 17.7 [14.1 to 21.4]
Statistical Analysis 1: Comparison: Carboplatin + Paclitaxel + Pembrolizumab + Olaparib vs Carboplatin + Paclitaxel; Test type: Superiority; p < 0.0001, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.51 to 0.79] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Carboplatin + Paclitaxel + Pembrolizumab vs Carboplatin + Paclitaxel; Test type: Superiority; p = 0.0981, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.70 to 1.08] — [estimate comment as in outcome 1, analysis 1]

14. Secondary Outcome: Time to First Subsequent Anti-cancer Treatment (TFST) in All Participants
Description: as for outcome 13
Time Frame: Up to approximately 67 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Carboplatin + Paclitaxel + Pembrolizumab + Olaparib | Carboplatin + Paclitaxel + Pembrolizumab | Carboplatin + Paclitaxel
Number analyzed (Participants) | 455 | 458 | 454
Months | 24.9 [22.0 to 29.5] | 18.2 [16.8 to 21.0] | 17.2 [15.3 to 19.0]
Statistical Analysis 1: Comparison: Carboplatin + Paclitaxel + Pembrolizumab + Olaparib vs Carboplatin + Paclitaxel; Test type: Superiority; p < 0.0001, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.59 to 0.80] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Carboplatin + Paclitaxel + Pembrolizumab vs Carboplatin + Paclitaxel; Test type: Superiority; p = 0.1206, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.79 to 1.06] — [estimate comment as in outcome 2, analysis 1]

15. Secondary Outcome: Time to Second Subsequent Anti-cancer Treatment (TSST) in Participants With PD-L1 Positive Tumors (CPS≥10)
Description: TSST is defined as the time from randomization to initiation of second subsequent anti-cancer treatment or death due to any cause, whichever occurs first. The TSST was determined from the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to approximately 67 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Carboplatin + Paclitaxel + Pembrolizumab + Olaparib | Carboplatin + Paclitaxel + Pembrolizumab | Carboplatin + Paclitaxel
Number analyzed (Participants) | 229 | 230 | 228
Months | 43.9 [33.5 to 52.5] | 36.3 [31.9 to 42.8] | 32.3 [27.5 to 39.2]
Statistical Analysis 1: Comparison: Carboplatin + Paclitaxel + Pembrolizumab + Olaparib vs Carboplatin + Paclitaxel; Test type: Superiority; p = 0.0316, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.80, 95% CI [0.63 to 1.01] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Carboplatin + Paclitaxel + Pembrolizumab vs Carboplatin + Paclitaxel; Test type: Superiority; p = 0.4441, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.98, 95% CI [0.78 to 1.24] — [estimate comment as in outcome 1, analysis 1]

16. Secondary Outcome: Time to Second Subsequent Anti-cancer Treatment (TSST) in All Participants
Description: as for outcome 15
Time Frame: Up to approximately 67 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Carboplatin + Paclitaxel + Pembrolizumab + Olaparib | Carboplatin + Paclitaxel + Pembrolizumab | Carboplatin + Paclitaxel
Number analyzed (Participants) | 455 | 458 | 454
Months | 34.7 [31.3 to 40.4] | 31.3 [28.1 to 34.2] | 30.9 [27.2 to 35.1]
Statistical Analysis 1: Comparison: Carboplatin + Paclitaxel + Pembrolizumab + Olaparib vs Carboplatin + Paclitaxel; Test type: Superiority; p = 0.0853, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.89, 95% CI [0.76 to 1.05] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Carboplatin + Paclitaxel + Pembrolizumab vs Carboplatin + Paclitaxel; Test type: Superiority; p = 0.7165, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.05, 95% CI [0.89 to 1.23] — [estimate comment as in outcome 2, analysis 1]

17. Secondary Outcome: Time to Discontinuation of Study Treatment or Death (TDT) in Participants With PD-L1 Positive Tumors (CPS≥10)
Description: TDT is defined as the time from the date of randomization to discontinuation of study treatment or death due to any cause, whichever occurs first. The TDT was determined from the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to approximately 67 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Carboplatin + Paclitaxel + Pembrolizumab + Olaparib | Carboplatin + Paclitaxel + Pembrolizumab | Carboplatin + Paclitaxel
Number analyzed (Participants) | 229 | 230 | 228
Months | 18.9 [14.9 to 22.4] | 15.3 [12.6 to 17.3] | 15.3 [13.0 to 17.3]
Statistical Analysis 1: Comparison: Carboplatin + Paclitaxel + Pembrolizumab + Olaparib vs Carboplatin + Paclitaxel; Test type: Superiority; p = 0.1029, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.71 to 1.08] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Carboplatin + Paclitaxel + Pembrolizumab vs Carboplatin + Paclitaxel; Test type: Superiority; p = 0.8231, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.90 to 1.36] — [estimate comment as in outcome 1, analysis 1]

18. Secondary Outcome: Time to Discontinuation of Study Treatment or Death (TDT) in All Participants
Description: as for outcome 17
Time Frame: Up to approximately 67 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Carboplatin + Paclitaxel + Pembrolizumab + Olaparib | Carboplatin + Paclitaxel + Pembrolizumab | Carboplatin + Paclitaxel
Number analyzed (Participants) | 455 | 458 | 454
Months | 17.7 [15.7 to 19.5] | 14.1 [12.4 to 15.4] | 15.2 [13.6 to 16.6]
Statistical Analysis 1: Comparison: Carboplatin + Paclitaxel + Pembrolizumab + Olaparib vs Carboplatin + Paclitaxel; Test type: Superiority; p = 0.0442, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.88, 95% CI [0.76 to 1.02] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Carboplatin + Paclitaxel + Pembrolizumab vs Carboplatin + Paclitaxel; Test type: Superiority; p = 0.9565, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.14, 95% CI [0.98 to 1.31] — [estimate comment as in outcome 2, analysis 1]

19. Secondary Outcome: Pathological Complete Response (pCR) Rate in Participants With PD-L1 Positive Tumors (CPS≥10)
Description: pCR is defined as the disappearance of all known disease noted prior to surgery; all surgical specimens collected during the interval debulking surgery are microscopically negative for malignancy. The percentage of participants who experience pCR was determined based on Miettinen & Nurminen method stratified by Bevacizumab use (yes versus no).
Time Frame: Up to approximately 21 months
Population: The analysis population includes all randomized participants with CPS≥10 who had pCR evaluation. Participants were analyzed in the treatment group to which they were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Pooled Carboplatin+Paclitaxel+Pembrolizumab+Olaparib, and Carboplatin+Paclitaxel+Pembrolizumab: This arm represents all participants who received pembrolizumab, per the pre-specified statistical analysis plan. Participants received carboplatin/paclitaxel via intravenous (IV) infusion for five 3-week cycles PLUS pembrolizumab 200 mg via IV infusion on Day 1 of each 3-week cycle for up to 35 cycles PLUS EITHER olaparib 300 mg OR placebo for olaparib via oral tablet twice each day (BID), starting with Cycle 7. Participants who experience severe hypersensitivity reaction to paclitaxel or an AE requiring discontinuation of paclitaxel may receive docetaxel (75 mg/m^2 Q3W) plus carboplatin AUC 5 Q3W after Sponsor consultation. Participants may also receive bevacizumab via IV infusion on Day 1 of each 3-week cycle at the Investigator's discretion.
Arm/Group | Pooled Carboplatin+Paclitaxel+Pembrolizumab+Olaparib, and Carboplatin+Paclitaxel+Pembrolizumab | Carboplatin + Paclitaxel
Number analyzed (Participants) | 174 | 89
Percentage of Participants | 9.8 [5.8 to 15.2] | 4.5 [1.2 to 11.1]
Statistical Analysis 1: Comparison: Pooled Carboplatin+Paclitaxel+Pembrolizumab+Olaparib, and Carboplatin+Paclitaxel+Pembrolizumab vs Carboplatin + Paclitaxel; Test type: Superiority; p = 0.0644, t-test, 1 sided — One-sided p-value for testing. H0: difference in % = 0 versus H1: difference in % > 0; Difference in Percentage = 5.4, 95% CI 2-sided [-1.9 to 11.5] — Based on Miettinen & Nurminen method stratified by bevacizumab use (Yes vs No)

20. Secondary Outcome: Pathological Complete Response (pCR) Rate in All Participants
Description: pCR is defined as the disappearance of all known disease noted prior to surgery; all surgical specimens collected during the interval debulking surgery are microscopically negative for malignancy. The percentage of participants who experience pCR was determined based on Miettinen & Nurminen method stratified by Bevacizumab use (yes versus no) and PD-L1 status (CPS <10 versus CPS>=10).
Time Frame: Up to approximately 26 months
Population: The analysis population includes all randomized participants who had pCR evaluation. Participants were analyzed in the treatment group to which they were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pooled Carboplatin+Paclitaxel+Pembrolizumab+Olaparib, and Carboplatin+Paclitaxel+Pembrolizumab | Carboplatin + Paclitaxel
Number analyzed (Participants) | 339 | 171
Percentage of Participants | 5.9 [3.6 to 9.0] | 2.3 [0.6 to 5.9]
Statistical Analysis 1: Comparison: Pooled Carboplatin+Paclitaxel+Pembrolizumab+Olaparib, and Carboplatin+Paclitaxel+Pembrolizumab vs Carboplatin + Paclitaxel; Test type: Superiority; p = 0.0318, t-test, 1 sided — One-sided p-value for testing. H0: difference in % = 0 versus H1: difference in % > 0; Difference in Percentage = 3.7, 95% CI 2-sided [-0.3 to 7.3] — Based on Miettinen & Nurminen method stratified by bevacizumab use (Yes vs No) and PD-L1 CPS (<10 vs ≥10)

21. Secondary Outcome: Number of Participants Who Experience an Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience an AE will be reported.
Time Frame: Up to approximately 73 months (anticipated)
Reporting Status: Not Posted, anticipated posting 2027-05

22. Secondary Outcome: Number of Participants Who Discontinue Study Treatment Due to an AE
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study intervention due to an AE will be reported.
Time Frame: Up to approximately 6 years (anticipated)
Reporting Status: Not Posted, anticipated posting 2027-05

ADVERSE EVENTS:
Time Frame: Up to approximately 67 months
Description: The population for all-cause mortality includes all participants. AE populations include all randomized participants who received at least 1 dose of study drug. Terms 'Neoplasm progression' 'Malignant neoplasm progression' and 'Disease progression' not related to the drug are excluded.
Arm/Group | Carboplatin + Paclitaxel + Pembrolizumab + Olaparib | Carboplatin + Paclitaxel + Pembrolizumab | Carboplatin + Paclitaxel
All-Cause Mortality (participants affected / at risk) | 237/455 | 243/458 | 229/454
Serious Adverse Events (participants affected / at risk) | 205/452 | 179/456 | 122/454
Other Adverse Events (participants affected / at risk) | 445/452 | 442/456 | 445/454
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carboplatin + Paclitaxel + Pembrolizumab + Olaparib (N=452) | Carboplatin + Paclitaxel + Pembrolizumab (N=456) | Carboplatin + Paclitaxel (N=454)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 5 (5) | 4 (4)
Aplasia pure red cell (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 19 (19) | 16 (17) | 9 (11)
Leukopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 1 (1)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 5 (5) | 3 (3) | 3 (3)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0)
Autoimmune myocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Bundle branch block left (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2) | 2 (2)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular hypokinesia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 4 (4) | 4 (4) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 2 (2) | 2 (2) | 0 (0)
Hypopituitarism (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0)
Thyroid disorder (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Thyroiditis (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0)
Macular hole (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vogt-Koyanagi-Harada disease (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal adhesions (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 1 (1) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 4 (4) | 2 (2)
Colitis (Gastrointestinal disorders) | 4 (4) | 6 (7) | 2 (2)
Colonic fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (6) | 2 (3) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Enterocutaneous fistula (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 5 (5) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Hernial eventration (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Ileal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 6 (6) | 6 (8) | 4 (4)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 8 (11) | 9 (10) | 6 (6)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Large intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (4) | 1 (1) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatic cyst (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatic fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 7 (8) | 7 (8) | 7 (11)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (5) | 3 (3) | 1 (1)
Administration site extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 2 (2) | 1 (1) | 2 (2)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 2 (2) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (2)
General physical health deterioration (General disorders) | 2 (3) | 1 (1) | 2 (2)
Hernia (General disorders) | 2 (2) | 1 (1) | 1 (1)
Hyperpyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Ill-defined disorder (General disorders) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1) | 1 (2)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Performance status decreased (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 15 (18) | 7 (9) | 4 (4)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0) | 1 (1)
Vaccination site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Biliary fistula (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholangitis sclerosing (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic cytolysis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 1 (1) | 0 (0)
Hepatic haemorrhage (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic necrosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatitis toxic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatobiliary disease (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (2)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 2 (2) | 0 (0)
Contrast media allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 1 (3) | 0 (0)
Eosinophilic granulomatosis with polyangiitis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 2 (2) | 1 (1)
Type IV hypersensitivity reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Abdominal infection (Infections and infestations) | 0 (0) | 3 (4) | 0 (0)
Acid fast bacilli infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacterial pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Biloma infected (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 9 (9) | 2 (2) | 3 (4)
COVID-19 pneumonia (Infections and infestations) | 6 (6) | 4 (4) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Colostomy infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 4 (4) | 3 (4) | 1 (1)
Device related sepsis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Encephalitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Enterocolitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Hepatitis E (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Infected cyst (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infected lymphocele (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Infected seroma (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Klebsiella infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Malaria (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Mastitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pelvic abscess (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Periodontitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Perirectal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 7 (9) | 8 (8) | 1 (1)
Pneumonia aspiration (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 2 (3) | 2 (2) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Rhinovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 3 (3) | 5 (5)
Septic shock (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 14 (17) | 7 (7) | 9 (10)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Anastomotic complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Anastomotic stenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Chemical peritonitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal stoma necrosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Post procedural fistula (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Wound evisceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (3) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Coagulation factor decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 4 (4) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4) | 4 (4) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Endocrine neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Endometrial stromal sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Intraductal papilloma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Uterine carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
IIIrd nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Meningitis noninfective (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Motor neurone disease (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Partial seizures (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 2 (3) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 5 (7) | 3 (3) | 1 (1)
Bladder perforation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 1 (1)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 3 (4)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 4 (4) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Immune-mediated dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Euthanasia (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Arterial thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphocele (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Vasculitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carboplatin + Paclitaxel + Pembrolizumab + Olaparib (N=452) | Carboplatin + Paclitaxel + Pembrolizumab (N=456) | Carboplatin + Paclitaxel (N=454)
Anaemia (Blood and lymphatic system disorders) | 270 (488) | 212 (344) | 205 (322)
Leukopenia (Blood and lymphatic system disorders) | 90 (201) | 60 (110) | 60 (113)
Neutropenia (Blood and lymphatic system disorders) | 170 (437) | 138 (309) | 147 (317)
Thrombocytopenia (Blood and lymphatic system disorders) | 89 (180) | 73 (127) | 72 (127)
Hyperthyroidism (Endocrine disorders) | 33 (37) | 44 (49) | 23 (25)
Hypothyroidism (Endocrine disorders) | 89 (107) | 93 (111) | 42 (50)
Abdominal distension (Gastrointestinal disorders) | 26 (28) | 26 (28) | 24 (29)
Abdominal pain (Gastrointestinal disorders) | 91 (133) | 90 (114) | 102 (143)
Abdominal pain upper (Gastrointestinal disorders) | 50 (70) | 54 (67) | 42 (49)
Constipation (Gastrointestinal disorders) | 121 (166) | 122 (147) | 104 (137)
Diarrhoea (Gastrointestinal disorders) | 121 (194) | 138 (247) | 94 (149)
Dyspepsia (Gastrointestinal disorders) | 40 (44) | 22 (25) | 28 (31)
Nausea (Gastrointestinal disorders) | 227 (432) | 187 (321) | 150 (262)
Stomatitis (Gastrointestinal disorders) | 46 (52) | 35 (41) | 30 (45)
Vomiting (Gastrointestinal disorders) | 114 (172) | 81 (120) | 70 (94)
Asthenia (General disorders) | 116 (176) | 97 (158) | 70 (108)
Fatigue (General disorders) | 120 (159) | 115 (179) | 85 (118)
Mucosal inflammation (General disorders) | 33 (41) | 23 (30) | 17 (23)
Oedema peripheral (General disorders) | 35 (39) | 28 (33) | 36 (50)
Pyrexia (General disorders) | 66 (85) | 50 (65) | 34 (42)
COVID-19 (Infections and infestations) | 65 (70) | 53 (57) | 53 (53)
Cystitis (Infections and infestations) | 24 (41) | 15 (20) | 14 (19)
Nasopharyngitis (Infections and infestations) | 21 (27) | 26 (34) | 30 (48)
Urinary tract infection (Infections and infestations) | 91 (151) | 79 (130) | 85 (144)
Alanine aminotransferase increased (Investigations) | 74 (114) | 65 (102) | 71 (115)
Aspartate aminotransferase increased (Investigations) | 68 (110) | 64 (112) | 59 (109)
Blood alkaline phosphatase increased (Investigations) | 26 (35) | 33 (55) | 22 (38)
Blood creatinine increased (Investigations) | 46 (92) | 21 (27) | 22 (30)
Lymphocyte count decreased (Investigations) | 28 (61) | 19 (49) | 7 (21)
Neutrophil count decreased (Investigations) | 104 (336) | 96 (236) | 102 (244)
Platelet count decreased (Investigations) | 79 (133) | 65 (117) | 58 (107)
Weight decreased (Investigations) | 51 (54) | 37 (38) | 28 (28)
Weight increased (Investigations) | 12 (14) | 23 (24) | 18 (20)
White blood cell count decreased (Investigations) | 88 (254) | 63 (154) | 80 (187)
Decreased appetite (Metabolism and nutrition disorders) | 83 (105) | 69 (88) | 52 (63)
Hyperglycaemia (Metabolism and nutrition disorders) | 23 (38) | 18 (21) | 20 (30)
Hypokalaemia (Metabolism and nutrition disorders) | 43 (78) | 44 (55) | 21 (34)
Hypomagnesaemia (Metabolism and nutrition disorders) | 49 (81) | 53 (81) | 58 (98)
Hyponatraemia (Metabolism and nutrition disorders) | 24 (39) | 23 (35) | 20 (30)
Arthralgia (Musculoskeletal and connective tissue disorders) | 136 (211) | 142 (243) | 139 (229)
Back pain (Musculoskeletal and connective tissue disorders) | 63 (77) | 48 (55) | 67 (76)
Bone pain (Musculoskeletal and connective tissue disorders) | 20 (33) | 13 (16) | 23 (33)
Myalgia (Musculoskeletal and connective tissue disorders) | 72 (104) | 82 (124) | 75 (98)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 38 (58) | 61 (79) | 45 (65)
Dizziness (Nervous system disorders) | 52 (63) | 41 (57) | 43 (58)
Dysgeusia (Nervous system disorders) | 41 (51) | 35 (36) | 22 (30)
Headache (Nervous system disorders) | 87 (119) | 67 (103) | 77 (115)
Hypoaesthesia (Nervous system disorders) | 23 (35) | 18 (31) | 22 (31)
Neuropathy peripheral (Nervous system disorders) | 85 (93) | 91 (101) | 83 (96)
Paraesthesia (Nervous system disorders) | 32 (38) | 32 (33) | 35 (44)
Peripheral sensory neuropathy (Nervous system disorders) | 54 (71) | 68 (77) | 56 (65)
Anxiety (Psychiatric disorders) | 19 (20) | 21 (22) | 23 (24)
Insomnia (Psychiatric disorders) | 35 (45) | 38 (45) | 45 (51)
Dysuria (Renal and urinary disorders) | 29 (31) | 11 (11) | 17 (24)
Proteinuria (Renal and urinary disorders) | 33 (56) | 36 (50) | 37 (44)
Cough (Respiratory, thoracic and mediastinal disorders) | 46 (49) | 46 (54) | 41 (54)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 55 (65) | 51 (61) | 41 (50)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 38 (47) | 38 (54) | 47 (67)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 30 (32) | 17 (20) | 26 (30)
Alopecia (Skin and subcutaneous tissue disorders) | 123 (125) | 114 (115) | 131 (131)
Pruritus (Skin and subcutaneous tissue disorders) | 63 (82) | 69 (95) | 57 (74)
Rash (Skin and subcutaneous tissue disorders) | 69 (88) | 71 (92) | 42 (51)
Hot flush (Vascular disorders) | 18 (23) | 23 (25) | 29 (33)
Hypertension (Vascular disorders) | 52 (60) | 76 (99) | 76 (103)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (2):
  • Study Protocol (2025-08-19): https://cdn.clinicaltrials.gov/large-docs/65/NCT03740165/Prot_001.pdf
  • Statistical Analysis Plan (2023-01-05): https://cdn.clinicaltrials.gov/large-docs/65/NCT03740165/SAP_002.pdf